CLINICAL TRIAL: NCT02187939
Title: Get in the GROOVE (Girls Realizing Options Through OpenSim Virtual Experiences)!
Brief Title: Get in the GROOVE!
Acronym: GROOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Patricia and Phillip Frost Museum of Science (formerly known as Miami Science Museum) (Unknown); New York Hall of Science (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Patrice G. Saab, Principal Investigator; Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20111081; 5R25OD010525 (NIH)
Record Dates: First submitted 2014-06-30; First posted 2014-07-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Health Behavior; Prevention Harmful Effects
MeSH Terms: conditions — Health Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Summer wellness program - nutrition & physical activity (Active Comparator): The GROOVE condition uses conventional means to address health-related activities and content within the context of a science museum summer enrichment program. The emphasis is on nutrition, physical activity, and healthy lifestyle.
  Interventions: Other: Summer science wellness program emphasizing health education pertaining to nutrition, physical activity, and healthy lifestyle.
- Summer program plus virtual world technology (Experimental): The GROOVE+ condition enhances the conventional approach to address health-related activities and content within the context of a science museum summer enrichment program by employing technology and a 3-D virtual world as a key educational strategy. The emphasis is on nutrition, physical activity, and healthy lifestyle.
  Interventions: Other: Summer science wellness program emphasizing health education pertaining to nutrition, physical activity, and healthy lifestyle.

INTERVENTIONS:
Other: Summer science wellness program emphasizing health education pertaining to nutrition, physical activity, and healthy lifestyle. — The enhanced virtual world education (GROOVE+) will be compared to conventional approach (GROOVE). Each program is Monday-Friday, 9:30-3:30, for 3 weeks in the summer.

SUMMARY:
Get in the GROOVE! will address health disparities impacting underserved youth. Given the alarming rate of overweight and obesity among high school minority youth, the project will focus on middle school with the primary aim of reaching middle school girls before unhealthy habits become firmly ingrained.

The primary aim of the research project is to investigate the impact of two types of summer science enrichment programs (that focus on health and wellness) on middle school girls' self-efficacy, health knowledge, health behaviors, and interest in science. One program will present the curriculum by conventional means (GROOVE condition) while the second program will include the addition of a closed 3-D virtual world environment to reinforce concepts (GROOVE+ condition).

The following hypotheses will be tested in the randomized controlled trial:

1. Upon completion of the summer program, the enhanced summer program GROOVE+ relative to the conventional summer program will result in a) increased self-efficacy for adopting healthy behavior change; b) increased health knowledge; c) enhanced science self-concept; and e) more positive behavior change (e.g., improved nutrition, increased physical activity).
2. At follow-up, the enhanced summer program relative to the conventional summer program will result in further and/or sustained improvements in positive behavior health behaviors and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Girls 11-14 years old

Exclusion Criteria:

Girls are excluded if they are:

* not fluent in English
* enrolled in a special education program at school (other than gifted program) that would interfere with ability to master the material
* have a condition that would preclude their participation in the dance activities of the summer program

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
change in Health Knowledge | pretreatment ( Day1-2) and post treatment (end of 3 week summer session)
  Multiple choice questionnaire used to assess participants' health knowledge pertaining to nutrition, physical activity, weight, and lifestyle. The measure will test for the content of the summer program.

SECONDARY OUTCOMES:
change in Self-efficacy - physical activity | pretreatment ( Day1-2) and post treatment (end of 3 week summer session)
  The physical activity self-efficacy support seeking and barriers subscales developed by Saunders, Pate, Felton et al.'s (1997, Preventive Medicine, vol. 26, 241-247) will be used.
change in Self-efficacy - fruit and vegetable consumption | pretreatment ( Day1-2) and post treatment (end of 3 week summer session)
  The food-related self-efficacy scale items comes from the work of Reynolds et al. ( 2002, Health Psychology, vol. 21, 51-60) and addresses fruit and vegetable consumption.
change in Self-efficacy - science | pretreatment ( Day1-2) and post treatment (end of 3 week summer session)
  Science self-efficacy assesses confidence to master the GROOVE program science components.

OTHER OUTCOMES:
change in health behaviors | pretreatment ( Day1-2), post treatment (end of 3 week summer session), and up to a year follow-up
  eating habits and physical activity habits
change in Science attitudes and aspirations | pretreatment ( Day1-2), post treatment (end of 3 week summer session), and up to a year follow-up
  This measure consist of items drawn from Louise Archer et al.'s (2013, Journal of Education Policy, 1-28, http://www.tandfonline.com/doi/abs/10.1080/02680939.2013.790079#.UbDmUuARtm1) ASPIRES project. Participants are asked to make ratings reflecting science attitudes, aspirations, and interests.
change in Family and participant habits | pretreatment ( Day1-2), post treatment (end of 3 week summer session - for participant only), and up to a year follow-up
  Assesses family and participant activities and habits and ratings of participant health and interests.
change in Pedometer activity | Participants will be given a pedometer to wear during the 3 week summer program period
  Pedometers will be used daily to assess physical activity.
Change in eating behavior | Up to 4 assessments will occur over the 3 week program.
  The Eating Behavior Scale consists of 28 items; all 20 items from Fahlman et al. (2013, American Journal of Health Education, vol. 43, 165-171) and 8 additional items from the 2009-2010 School Physical Activity and Nutrition Project (https://sph.uth.edu/content/uploads/2011/12/SPAN_2009-10_8th-11thStudentSurveyEnglish_FINAL.pdf). The measure asks participants to indicate how many times they consumed an item on the day before (e.g., fruits, vegetables, candy, etc). A subsample of students will complete up to three 24-hour dietary recalls to examine the validity of the self-report items in the study's participants.
change in Presence | up to 3 times during the GROOVE+ condition
  The presence scale consists of 11 items influenced by the work of Fox et al. (2009, Presence Vol. 18,294-303) will be completed by the participants in the GROOVE+ condition. The scale assesses the extent to which the participant feels present in the 3-D virtual world.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice G Saab, Ph.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Patricia and Phillip Museum of Science, Miami, Florida
  - New York Hall of Science, Queens, New York